CLINICAL TRIAL: NCT03819088
Title: Effects on QOL When Zinc is Supplemented in Patients With Upper GI Cancer on Chemotherapy
Brief Title: Effects on Quality of Life With Zinc Supplementation in Patients With Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00099791; NCI-2017-02467 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4173-17 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Gastric Carcinoma; Liver and Intrahepatic Bile Duct Carcinoma; Unresectable Esophageal Carcinoma; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (zinc months 1 and 2) (Experimental): Patients receive zinc PO TID for months 1 and 2 only of the first 4 months on therapy.
  Interventions: Dietary Supplement: Zinc
- Group II (zinc months 3 and 4) (Experimental): Patients receive zinc PO TID for months 3 and 4 only of the first 4 months on therapy.
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — Given PO
  Other Names: Zinc sulfate

SUMMARY:
This randomized study examines how well zinc works in improving quality of life in patients with gastrointestinal cancer that cannot be removed by surgery who are receiving chemotherapy. Zinc may help to improve patient's quality of life by preventing zinc deficiency.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the effects on quality of life (QOL) when supplementing zinc in upper gastrointestinal (GI) cancer patients while they are receiving chemotherapy.

SECONDARY OBJECTIVES:

I. Correlate hypoalbuminemia with serum zinc deficiency.

II. Correlate zinc deficiency with neutropenia.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive zinc orally (PO) thrice daily (TID) for months 1 and 2 only of the first 4 months on therapy.

GROUP II: Patients receive zinc orally (PO) TID for months 3 and 4 only of the first 4 months on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to adult medical oncology outpatient clinic with new diagnosis of non-resectable gastric, gastro-esophageal, pancreas or biliary cancer
* Patients plan to receive chemotherapy at an Emory Cancer Center
* No prior chemotherapy or radiation therapy for newly diagnosed gastric, gastro-esophageal, pancreas or biliary cancer
* Patients must sign informed consent

Exclusion Criteria:

* Zinc supplementation is not indicated for pregnant or lactating women therefore, this is an exclusion criteria and women of childbearing age will complete a pregnancy test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Quality of life scores | Up to 4 months after study start
  Quality of life (QOL) will be evaluated through patient subjective responses to the QOL survey.

SECONDARY OUTCOMES:
Serum zinc level | Up to 4 months after study start
  Zinc levels will be monitored monthly with blood tests. Low zinc will be defined as under 60 mcg.
Serum albumin level | Up to 4 months after study start
  Albumin levels will be monitored monthly with blood tests. Low albumin will be defined as under 3.5 gm/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji B. Alese, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
Plan may be reevaluated at the time of publication.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT03819088/ICF_000.pdf